CLINICAL TRIAL: NCT04369950
Title: Post-cesarean Analgesia With Epidural Morphine Following Epidural 2-chloroprocaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Linden Lee, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-19-0951
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Results first posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-04

CONDITIONS: Physiological Effect of Drugs; Morphine; Analgesics; Analgesics, Opioid; Central Nervous System Depressants; Narcotics
Keywords: cesarean delivery; c-section; chloroprocaine; lidocaine; morphine; post-operative pain; post-cesarean analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine; Epinephrine; chloroprocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2 percent Lidocaine with epinephrine and epidural morphine (Active Comparator)
  Interventions: Drug: 2% lidocaine with 1:200,000 epinephrine and epidural morphine
- 3 percent 2-Chloroprocaine and epidural morphine (Experimental)
  Interventions: Drug: 3% 2-chloroprocaine and epidural morphine

INTERVENTIONS:
Drug: 2% lidocaine with 1:200,000 epinephrine and epidural morphine — Epidurals will be dosed with 2% lidocaine with 1:200,000 epinephrine to T4 level in 5ml increments, epidural morphine 3mg will be given after delivery of neonate. T4 level maintained throughout cesarean delivery with additional epidural doses of 2% lidocaine with 1:200,000 epinephrine for both groups. Post-operative orders of scheduled acetaminophen and ibuprofen, and oxycodone as needed will be written.
  Arms: 2 percent Lidocaine with epinephrine and epidural morphine
Drug: 3% 2-chloroprocaine and epidural morphine — Epidurals will be dosed with 3% 2-chloroprocaine to T4 level in 5ml increments, epidural morphine 3mg will be given after delivery of neonate. T4 level maintained throughout cesarean delivery with additional epidural doses of 2% lidocaine with 1:200,000 epinephrine for both groups. This is the critical component to bridge the latency period between the offset of 3% 2-chloroprocaine and the peak action of epidural morphine.Post-operative orders of scheduled acetaminophen and ibuprofen, and oxycodone as needed will be written.
  Arms: 3 percent 2-Chloroprocaine and epidural morphine

SUMMARY:
The purpose of this study is to show that the effect of 3% 2-chloroprocaine prior to epidural morphine administration will be not inferior to the effect of epidural 2% lidocaine with 1:200,000 epinephrine on total opioid use for 24h

ELIGIBILITY:
Inclusion Criteria:

* pregnant patients
* live singleton pregnancy

Exclusion Criteria:

* BMI >40
* obstructive sleep apnea
* drug abuse
* chronic pain
* chronic opioid use
* nonfunctioning epidural

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linden Lee, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee LO, Ramirez-Chapman AL, White DL, Zhang X, Lu M, Suresh MS. Postcesarean Analgesia With Epidural Morphine After Epidural 2-Chloroprocaine: A Randomized Noninferiority Trial. Anesth Analg. 2023 Jan 1;136(1):86-93. doi: 10.1213/ANE.0000000000006109. Epub 2022 Jun 3. PMID 36534717

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 2 Percent Lidocaine With Epinephrine and Epidural Morphine | 3 Percent 2-Chloroprocaine and Epidural Morphine
Started | 22 | 22
Completed | 20 | 20
Not Completed | 2 | 2
Not completed — Protocol Violation | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 Percent Lidocaine With Epinephrine and Epidural Morphine | 3 Percent 2-Chloroprocaine and Epidural Morphine | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (5.4) | 29.8 (5.4) | 28.7 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 8 | 8 | 16
  Hispanic | 7 | 5 | 12
  Caucasian | 4 | 5 | 9
  Asian | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Height [Mean (Standard Deviation); unit: centimeters] | 159.5 (6.9) | 163 (7.5) | 161.25 (7.20)
Weight [Mean (Standard Deviation); unit: kilograms] | 84.0 (13.2) | 87.1 (14.8) | 85.55 (14.02)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.3 (4.4) | 32.4 (4.2) | 32.35 (4.30)
Number of Participants who Smoke [Count of Participants; unit: Participants] | 0 | 0 | 0
Gestational age [Mean (Standard Deviation); unit: weeks] | 38.7 (1.1) | 38.6 (1.1) | 38.65 (1.1)
Gravida [Median (Inter-Quartile Range); unit: pregnancies] | 1 [1 to 1] | 2 [1 to 2] | 1 [1 to 2]
Para [Median (Inter-Quartile Range); unit: completed pregnancies] — number of completed pregnancies beyond 20 weeks gestation (whether viable or nonviable)
  completed pregnancies | 0 [0 to 0] | 0 [0 to 1] | 0 [0 to 1]
Duration of labor analgesia [Mean (Standard Deviation); unit: hours] | 8.5 (4.8) | 7.9 (5.6) | 8.2 (5.21)
Surgical duration [Median (Inter-Quartile Range); unit: minutes] | 34.5 [30 to 52] | 42 [35.5 to 57.5] | 38.5 [30.5 to 57]
Number of participants who received a labor analgesia with combined spinal epidural [Count of Participants; unit: Participants] | 3 | 2 | 5
Number of Participants with Prior Cesarean Delivery / trial of labor after cesarean [Count of Participants; unit: Participants] | 0 | 3 | 3
Surgical Complication (uterine artery laceration and postpartum hemorrhage) [Count of Participants; unit: Participants] | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Total Amount of Opioid Used
Time Frame: 24 hours after epidural morphine administration
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | 2 Percent Lidocaine With Epinephrine and Epidural Morphine | 3 Percent 2-Chloroprocaine and Epidural Morphine
Number analyzed (Participants) | 20 | 20
milligrams | 15 [6.3 to 22.5] | 0 [0 to 15.6]

2. Secondary Outcome: Total Amount of Opioid Used
Time Frame: 12 hours after epidural morphine administration
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | 2 Percent Lidocaine With Epinephrine and Epidural Morphine | 3 Percent 2-Chloroprocaine and Epidural Morphine
Number analyzed (Participants) | 20 | 20
hours | 0 [0 to 7.5] | 0 [0 to 10]

3. Secondary Outcome: Total Amount of Opioid Used
Time Frame: 8 hours after epidural morphine administration
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | 2 Percent Lidocaine With Epinephrine and Epidural Morphine | 3 Percent 2-Chloroprocaine and Epidural Morphine
Number analyzed (Participants) | 20 | 20
hours | 0 [0 to 7.5] | 0 [0 to 10]

4. Secondary Outcome: Total Amount of Opioid Used
Time Frame: 4 hours after epidural morphine administration
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | 2 Percent Lidocaine With Epinephrine and Epidural Morphine | 3 Percent 2-Chloroprocaine and Epidural Morphine
Number analyzed (Participants) | 20 | 20
hours | 0 [0 to 0] | 0 [0 to 8.1]

5. Secondary Outcome: Pain as Measured by a 11 Point Verbal Scale
Description: scale ranges form 0-10, higher number indicating more pain
Time Frame: 4,8, 12 and 24 hours after epidural morphine administration
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 2 Percent Lidocaine With Epinephrine and Epidural Morphine | 3 Percent 2-Chloroprocaine and Epidural Morphine
Number analyzed (Participants) | 20 | 20
score on a scale
  4 hours | 0 [0 to 1] | 2.5 [0 to 5]
  8 hours | 0 [0 to 4.5] | 1 [0 to 4]
  12 hours | 3 [0 to 5] | 2 [0 to 3]
  24 hours | 7 [4 to 7.5] | 3.5 [1 to 6]

6. Secondary Outcome: Number of Participants Who Had Mild, Moderate or Severe Nausea as Measured by a 3 Point Scale
Description: scale ranges from non,mild and moderate-severe
Time Frame: 4,8, 12 and 24 hours after epidural morphine administration
Measure: Count of Participants; unit: Participants
Arm/Group | 2 Percent Lidocaine With Epinephrine and Epidural Morphine | 3 Percent 2-Chloroprocaine and Epidural Morphine
Number analyzed (Participants) | 20 | 20
Participants
  4 hours | 3 | 1
  8 hours | 1 | 2
  12 hours | 0 | 0
  24 hours | 0 | 0

7. Secondary Outcome: Number of Participants Who Had Mild, Moderate or Severe Pruritis as Measured by a 3 Point Scale
Description: scale ranges from non,mild and moderate-severe
Time Frame: 4,8, 12 and 24 hours after epidural morphine administration
Measure: Count of Participants; unit: Participants
Arm/Group | 2 Percent Lidocaine With Epinephrine and Epidural Morphine | 3 Percent 2-Chloroprocaine and Epidural Morphine
Number analyzed (Participants) | 20 | 20
Participants
  4 hours | 7 | 3
  8 hours | 6 | 4
  12 hours | 4 | 3
  24 hours | 2 | 0

8. Secondary Outcome: Time Until First Opioid Request
Time Frame: Up to 48 hours after epidural morphine administration
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | 2 Percent Lidocaine With Epinephrine and Epidural Morphine | 3 Percent 2-Chloroprocaine and Epidural Morphine
Number analyzed (Participants) | 20 | 20
hours | 14.8 [7.9 to 22.7] | 24.7 [2.7 to 36.6]

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | 2 Percent Lidocaine With Epinephrine and Epidural Morphine | 3 Percent 2-Chloroprocaine and Epidural Morphine
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 10/20 | 6/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2 Percent Lidocaine With Epinephrine and Epidural Morphine (N=20) | 3 Percent 2-Chloroprocaine and Epidural Morphine (N=20)
Nausea (General disorders) | 5 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 5

LIMITATIONS AND CAVEATS:
No prior studies investigating the technique studied in order to calculate study size; wide interindividual differences in pain; physician administering epidural medications not blinded; originally intended to recruit 80, but due to recruitment challenges decided to modify recruitment goal to about 40 and classify this as an exploratory study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/50/NCT04369950/Prot_SAP_000.pdf